CLINICAL TRIAL: NCT06533111
Title: Improving Surgical Patient Outcomes Through Implementation of a SemiStructured Intraoperative Anesthesia Handoff Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Aubrey Samost-Williams, Assistant Professor Non-Tenure Clinical, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSC-MS-24-0552; 1K12TR004908-01 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Post-operative Complications
Keywords: Intraoperative anesthesia handoffs

STUDY DESIGN:
Intervention Model Description: The non-cardiac adult operating rooms at Memorial Hermann Hospital are split into 2 floors, Sarofim 2 and Sarofim 3. These floors will be the unit of clustering. One floor will be randomized to the intervention arm and the other to the control arm. Every 4 weeks both floors will be re-randomized again to either arm for a total of 18 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epic Health Record semi-structured handoff cognitive aid (Experimental)
  Interventions: Other: Epic Health Record semi-structured handoff cognitive aid
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Epic Health Record semi-structured handoff cognitive aid — Epic Health Record cognitive aid will be used for intraoperative anesthesia handoff
  Arms: Epic Health Record semi-structured handoff cognitive aid
Other: Usual care — Epic Health Record cognitive aid will not be used for intraoperative anesthesia handoff
  Arms: Usual care

SUMMARY:
The purpose of this study is to assess the impact of a semi-structured intraoperative anesthesia handoff tool on patient outcomes and to assess the validity of the 5-Factor Perceived Shared Mental Model Scale (5-PSMMS) in a healthcare setting and whether the perception of Shared Mental Model (SMM) mediates the effect of the intraoperative handoff tool on postoperative outcomes

ELIGIBILITY:
Inclusion Criteria:

* Undergoing non-cardiac surgery in the main operating rooms (e.g. not the endoscopy suite or labor and delivery ward)
* Undergoing at least one permanent (e.g. end of shift) anesthesia clinician handoff

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status 6 (organ donors)

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have Myocardial Injury after Non-Cardiac Surgery/Myocardial Infarction | upto 30 days after surgery
Number of participants that have Acute Kidney Injury | from baseline upto 30 days after surgery
Number of participants that need Post-op blood transfusion | upto 24 hours after surgery
Number of participants that need Prolonged intubation | end of surgery(about 180 minutes after start of surgery)
Number of participants that have Pneumonia | within 30 days after surgery
Number of participants that need reintubation | within 24 hours after surgery
Number of participants that need Rapid Response Team Activation | within 24 hours after surgery
Number of participants that need Readmission | within 30 days after surgery
Number of participants that die after surgery | 30 days after surgery

SECONDARY OUTCOMES:
Number of participants that have Postoperative Hypotension | within 24 hours after surgery
Number of participants that have Hypoxia | within 2 hours after surgery
Number of participants that have Uncontrolled pain | within 2 hours after surgery
  Pain score average >/= 5 on a 10-point scale
Number of participants that have Intraoperative hypotension | at least 15 minutes intraoperatively following first intraoperative anesthesia handoff
  Mean Arterial Pressure < 65 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Aubrey Samost-Williams, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samost-Williams A, Green CE, Kao LS, Sridhar S, Sessler DI, Turan A, Thomas EJ. Assessing the impact of a semi-structured intraoperative anaesthesia handoff cognitive aid on surgical patient outcomes: study protocol for a cluster randomised trial. BMJ Open. 2025 Nov 4;15(11):e110401. doi: 10.1136/bmjopen-2025-110401. PMID 41248419